CLINICAL TRIAL: NCT01280630
Title: A Multicentre Retrospective Study to Understand Anti-thrombotic Treatment Patterns and Outcomes of Acute Coronary Syndrome (ACS) Patients in India
Brief Title: Multicentre Retrospective Study to Understand Anti-thrombotic Treatment Patterns and Outcomes of Acute Coronary Syndrome (ACS) Patients
Acronym: TRACE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-XXX-2010/1
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS: Acute coronary syndrome Retrospective Registry
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
TRACE is a Multicentre Retrospective Study planned to gather follow up data for a period of 1 year in order to understand anti-thrombotic management patterns and outcomes of Acute Coronary Syndrome patients in India.

This retrospective study is designed to provide a rapid and quick analysis of the existing database of ACS patients. So as to ensure quality check in the study, a pilot study will be conducted with around 500 patients at 10 centres across India and based on the meaningful results of the pilot study, full retrospective multi-centric study will be initiated at various selected centres across India. This study will use available registry data from a defined time period of Jan 2007-Dec 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the age of 18 years or older and hospitalized for ACS within the previous 3 years.
* Diagnosis of STEMI, NSTEMI or UA using Standard and Universal Definition of Myocardial Infarction

Exclusion Criteria:

* UA, STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or GI bleeding or post-PCI.
* UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACS patients admitted in tertiary care hospitals
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Anti thrombotic strategies used in ACS patients | Jan 2007-Dec 2009
Anti-thrombotic treatment strategies in a 'real-life' observational setting across different sites in India. | Jan 2007-Dec 2009

SECONDARY OUTCOMES:
ACS outcomes with respect to: -Revascularization -Angina/ Re-infarction -Cardiogenic shock/Heart failure/Cardiac arrest -Atrial fibrillation/flutter -Ventricular Fibrillation/ Sustained V Tachycardia -Stroke -Mortality -Bleeding | Jan 2007-Dec 2009

CONTACTS AND LOCATIONS:
Overall Officials: Paurus M Irani, MD, Study Director — AZ India; Dr Jamshed Dalal, Principal Investigator — Kokila Ben Dhirubhai Ambani Hospital; Dr Keyur Parikh, Principal Investigator — Heart Care Hospitals; Dr S S Ramesh, Principal Investigator — Bhagwan Mahaveer Jain Hear Centre; Dr Upendra Kaul, Principal Investigator — Escorts Hospitals
Locations (7):
- India (7):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Chennai, Tamil Nadu